CLINICAL TRIAL: NCT05539053
Title: Efficacy of N-acetylcysteine for the Prevention and Relief of Paclitaxel-induced Peripheral Neuropathy in Women With Ovarian, Tubal, and Peritoneal Cancer: an Open-label, Randomized Controlled Trial
Brief Title: Efficacy of NAC for the Prevention and Relief of PIPN in Women With Ovarian, Tubal, and Peritoneal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 65068
Record Dates: First submitted 2022-07-27; First posted 2022-09-14 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-02

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — poly(methyl methacrylate)-b-polycaprolactone-N-acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NAC short course (Experimental): patient received CMT(Paclitaxel) and NAC 2400 mg/day one week per each cycle of CMT
  Interventions: Drug: N Acetylcysteine A
- NAC long course (Experimental): patient received CMT(Paclitaxel) and NAC 2400 mg/day every day for 9 weeks
  Interventions: Drug: N Acetylcysteine B
- control (No Intervention): patient received CMT(Paclitaxel) only

INTERVENTIONS:
Drug: N Acetylcysteine A — paclitaxel + N-Acetylcysteine orally short course
  Arms: NAC short course
Drug: N Acetylcysteine B — paclitaxel +N Acetylcysteine orally long course
  Arms: NAC long course

SUMMARY:
Ovarian cancer is third most common gynecologic cancer in Thai woman, treatment including surgery followed by chemotherapy.

Patient usually received paclitaxel every 3 week for 6 cycles, paclitaxel induce peripheral neuropathy is common dose dependent side effect which can disturb quality of life, result in chemotherapy dose reduction or discontinuation leading to poor prognosis and decreased survival Mechanism of PIPN including inflammation, promotion of microtubule polymerization and inhibition of depolymerization, and oxidative stress N-acetylcysteine is acetylated form of l-cysteine, might reduce oxidative stress. NAC can restore glutathione level, which is potent natural antioxidant. NAC might reduce PIPN

DETAILED DESCRIPTION:
This study was designed to evaluate the effect of NAC on the incidence and severity of PIPN in woman with ovarian, tubal, and peritoneal cancer who treated with paclitaxel for 3 cycles. (PIPPN is developed after cumulative doses 250 mg/m2 or more) Patient in controlled group, received Paclitaxel only. Patient in intervention group divided to two groups. First group received NAC 2400 mg/day for one week after received Paclitaxel each cycle for 3 cycles. Second group received NAC 2400 mg/day for 9 weeks Evaluate incidence and severity of PIPN before start CMT, and every visit after received CMT each cycle using Common Terminology Criteria for Adverse Event (CTCAE) ver.5, Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx), and Patient Neurotoxicity Questionnaire (PNQ)

ELIGIBILITY:
Inclusion Criteria:

* Female patient aged 18 years old or more with ovarian, tubal, and peritoneal cancer who received Paclitaxel first course after surgery
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Normal laboratory testing
* hemoglobin ≥10 g/dL, leukocyte count ≥ 3,000/mL, absolute neutrophil count ≥1,500/mL, platelet count ≥100,000/mL
* Serum creatinine ≤1.5 mg/dL
* Bilirubin ≤1.5 upper limit of normal
* Alkaline phosphatase and serum glutamic oxaloacetate transaminase ≤3 upper limit of normal

Exclusion Criteria:

* Patient with symptoms of peripheral neuropathy before study
* Allergy to N-acetylcysteine
* Psychiatric disorders
* Pregnant woman
* History of treated with other chemotherapy or radiotherapy before study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Paclitaxel-induce peripheral neuropathy | Day 0 (before chemotherapy administration), at the end of cycle 1, at the end of cycle 2, and at the end of cycle 3 (each cycle is 21 days)
  Assessment of grade of peripheral neuropathy by CTCAE v.5.0

SECONDARY OUTCOMES:
Severity of paclitaxel-induce peripheral neuropathy | Day 0 (before chemotherapy administration), at the end of cycle 1, at the end of cycle 2, and at the end of cycle 3 (each cycle is 21 days)
  Assessment of severity of peripheral neuropathy by Patient Neurotoxicity Questionnaire (PNQ)
Quality of life associated paclitaxel-induce peripheral neuropathy | Day 0 (before chemotherapy administration), at the end of cycle 1, at the end of cycle 2, and at the end of cycle 3 (each cycle is 21 days)
  Assessment of quality of life using FACT/GOG-Ntx

OTHER OUTCOMES:
Side effects of NAC | At the end of cycle 1, at the end of cycle 2, and at the end of cycle 3 (each cycle is 21 days)
  Nausea, vomiting, diarrhea, abdominal discomfort, allergy

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided